CLINICAL TRIAL: NCT05340452
Title: An Open Label, Randomized, Two Way Cross Over, Two Period, Two Treatment, Two Sequence Bioequivalence Study of Klaribact (Clarithromycin) 125mg/5ml Suspension Compared With Klaricid (Clarithromycin) 125mg/5ml Suspension in 24 Healthy Adult Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Klaribact 125mg/5ml, Suspension
Acronym: BE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Collaborators: Merck (Pvt.) Limited, Pakistan (Unknown); Center for Bioequivalence Studies and Clinical Research (CBSCR), HEJ Research Institute of chemistry, University of Karachi (Unknown)
Responsible Party: Principal Investigator, Dr. Muhammad Raza Shah, Professor, University of Karachi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CB-009-CLA-2012/Protocol/1.0
Record Dates: First submitted 2022-04-15; First posted 2022-04-22 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Bioequivalence Study; macrolide antibiotic; Bioavailability comparison
MeSH Terms: interventions — Suspensions; Clarithromycin

STUDY DESIGN:
Intervention Model Description: An Open Label, Randomized, Two Way Cross Over, Two Period, Two Treatment, Two Sequence Bioequivalence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Single oral dose of 20 ml of Test (Klaribact 125mg/5ml Suspension) will be given with the aid of graduated cup.
  Interventions: Drug: Klaribact 125mg/5ml Suspension
- Reference Group (Active Comparator): Single oral dose of 20 ml of Reference (Klaricid 125mg/5ml Suspension) will be given to volunteers with the aid of graduated cup.
  Interventions: Drug: Klaricid 125mg/5ml Suspension

INTERVENTIONS:
Drug: Klaribact 125mg/5ml Suspension — one single 20 mL dose (500mg) of the test drug will be administered to the volunteers
  Arms: Test Group
Drug: Klaricid 125mg/5ml Suspension — one single 20 mL dose (500mg) of the Reference drug will be administered to the volunteers
  Arms: Reference Group

SUMMARY:
A two way crossover BE study will be performed to evaluate the comparative bioavailability of Klaribact (Clarithromycin 125 mg/5ml) suspension (Merck Pvt. Ltd, Pakistan) with Klaricid (Clarithromycin 125mg/5ml) suspension (Abbot Laboratories Pakistan Limited) at the clinical site (CBSCR), Karachi Pakistan.

DETAILED DESCRIPTION:
The Bioequivalence study of Klaribact Suspension will be conducted on 24 healthy participants. Finally selected subjects will be divided into two groups, Group A and Group B, with 12 subjects in each group. The study will be consisted of two periods, Period I and Period II, each comprising of 35 hours, 11 hours before and 24 hours after the drug administration. A washout period of 6 days will be provided between the two periods to ensure the absence of carry over effect. Each group (A & B) will be treated with either of the two sequences, TR or RT, in Period I and the sequence will be inter-changed in Period II. blood samples from each volunteer will be collected at specific time points to analyze plasma concentration of Clarithromycin.

ELIGIBILITY:
Inclusion Criteria:

* All subjects should be healthy and free from any epidemic, contagious or measurable disease (e.g. Malaria, Dengue)
* Age range for inclusion will be 18-50 year.
* BMI for all Subjects will be between 18.5-26.9 kg/m2.
* Participant capable of understanding the informed consent.
* Non Smokers, who have not smoked in last 3 months.
* Availability of a study volunteer for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.
* Medical history, physical examination and screening tests must fall in normal range, unless the investigator considers the abnormality to be clinically not significant.
* Clinical laboratory test results should be within a normal range.
* Participants (who can read and understand urdu) should be able to give informed consent, understand and sign the Informed Consent Form.
* Participants should have adequate organ function (i.e., kidney, liver and heart).
* Subjects with negative urine screen for drugs of abuse. All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical screening procedures and at each study period check-in.
* Subjects having negative alcohol breathe test. All subjects will have breath alcohol test as part of the clinical screening procedures and at each study period check-in.

Exclusion Criteria:

* Any active allergic disease or a history of any significant allergic disease (e.g. Rhinitis, dermatitis, asthma).
* Known hypersensitivity to Investigational drug(s) or related class of drug(s).
* Abnormal results of blood and urine tests conducted at screening unless the investigator considers an abnormality to be clinically irrelevant.
* Presence or history of cardiac (e.g. Myocardial Infarction, arrythmia), renal (e.g. renal insufficiency) , hepatic (e.g. hepatic impairment) , organ insufficiency, bone marrow disease, hematological abnormality (e.g. leukemia, anemia), photosensitivity, neurological disorders (e.g. Alzheimer's disease) or gastrointestinal disease known to interfere with the drug absorption, distribution, metabolism or elimination (e.g. dysphagia).
* History or presence of any musculo skeletal disease (e.g. Tendonitis).
* Subject has donated blood (450ml) within 12 weeks minimum preceding the study. 16
* Alcoholic or with a history of chronic alcohol intake or consumed alcohol or Gutka in last 3 months.
* Ingestion of OTC drug, within 14 days of drug administration (e.g. aspirin, ibuprofen).
* History of intake of any prescribed medicine (e.g. captopril, sumatriptan) during a period of 30 days, prior to drug administration day of study.
* Ingestion of investigational drug within 30 days, prior to investigational drug administration in the study.
* Consumption of xanthine-containing products, tobacco containing products or alcohol for within 48 hours prior to dosing. or consume juice of grape fruit for within 14 days prior to study.
* Ingestion of any known hepatic or renal clearance altering agents (e.g. erythromycin, cimetidine, barbiturates, phenothiazines, etc.) for a period of 30 days, prior to study initiation. Drug interaction section at 5.13 should be considered.
* Subjects with an uncontrolled medical condition (i.e., hypertension, cardiac arrhythmias, CHF) that places the patient at risk by participating in the study.
* Subjects with known HIV, hepatitis B or C infection or autoimmune diseases.
* History of drug exposure which, in the opinion of Investigator, amounts to drug abuse.
* Participation in other drug studies within three months prior to study initiation.
* Subjects with any physical/mental disability.
* Limited mental capacity to the extent that the subject is unable to provide legal consent and information regarding the side effects or tolerance of the study drug.
* Subject who is unable to or likely to be non-compliant with protocol requirements or restrictions.
* Pregnancy or breast feeding, women of child bearing age who are not using a recognized form of contraception for at least last 30 days or using hormonal contraception, are also excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06-29 (Actual); Primary Completion 2013-07-08 (Actual); Study Completion 2013-10-25 (Actual)

PRIMARY OUTCOMES:
maximum plasma concentration | up to 24 hours post dose
  maximum drug concentration in plasma after dose
Time to reach maximum plasma concentration | 0 to 24 hours post dose
  Time required for the drug to reach maximum plasma concentration
AUC | 0 to 24hours post dose
  Area under the time versus plasma drug concentration curve

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shah, PhD, Principal Investigator — Center for bio-equivalence studies and clinical research (CBSCR); Naghma R Hashmi, PhD, Principal Investigator — Center for bio-equivalence studies and clinical research
Locations (1):
- Center for Bioequivalence Studies and clinical research (CBSCR), ICCBS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will only be available to other researchers upon reasonable request to PI keeping the participants' confidentiality intact.